CLINICAL TRIAL: NCT04317287
Title: A Double-blind, Randomized, Placebo-controlled, Parallel Design Study to Evaluate the Effects of the Cardio Formulation on Oxidized LDL in Individuals Who Are Overweight to Mildly Obese and Otherwise Healthy
Brief Title: To Assess the Efficacy and Safety of the Cardio Formulation in Reducing Oxidized LDL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 Pandemic
Sponsor: Supplement Formulators, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CL099
Record Dates: First submitted 2020-03-19; First posted 2020-03-23 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Oxidized Low Density Lipoprotein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardio formulation (Experimental): Tomato-based formulation with dietary supplement
  Interventions: Dietary Supplement: Cardio formulation
- Placebo (Placebo Comparator): Placebo softgels
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cardio formulation — Tomato-based formulation with dietary supplement softgels
  Arms: Cardio formulation
Dietary Supplement: Placebo — Placebo softgels
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of the Cardio formulation in reducing oxidized LDL [(Ox LDL (low density lipoprotein)] in overweight to mildly obese generally healthy adults.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled, parallel design study to evaluate the effectiveness of the Cardio formulation in reducing oxidized LDL. Each subject will receive a specific dose of the study product to be taken with a meal daily preferably at the same time each day with water.

Participants will receive questionnaires, assessments, blood tests, vital signs and body composition analysis.

The primary objective is the evaluation of the change in Ox LDL in response to the Cardio formulation at Days 30 and 60 relative to baseline compared with placebo.

The secondary objective is the evaluation of the change in anthropometric measurements, clinical laboratory evaluations, and health survey scores in response to the Cardio formulation at Days 30 and Day 60 relative to baseline compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory, male or female, 40-75 years of age
2. A BMI of 25-34.9 and/or waist circumference > 40.0 inches in males and > 35.0 inches in females
3. Having a fasting LDL cholesterol level of >100- <189 mg/dL OR, total cholesterol level of > 200-< 239 mg/dL OR triglycerides level of > 150 mg/dl - < 199 mg/dl OR blood sugar level > 100 mg/dl - < 126 mg/dl based upon the screening laboratory results from the Complete Blood Count (CBC)/Chemistry profile
4. Generally healthy and having no significant difficulty with digestion or absorption of food
5. Has been generally weight stable for the past six months (+ 6 lbs.)
6. Willing and able to give written informed consent
7. Clearly understands the procedures and study requirements
8. Willing and able to comply with all study procedures, including following the recommendations to maintain their usual diet and regular activity, as per protocol
9. Able to communicate, including reading, in English
10. Have not taken any nutritional supplements that may contain any of the components of the study product for a minimum of 14 days before Screening/baseline

Exclusion Criteria:

1. Having smoked any cigarette, electronic cigarette, cigar, pipe, or used a recreational drug or any product containing cannabidiol (CBD) or tetrahydrocannabinol (THC) in the past 30 days
2. Donated blood within 30 days before Screening/baseline
3. Inability to provide a venous blood sample
4. Participation in another study within 30 days prior to Screening/baseline
5. Being pregnant or planning on becoming pregnant during study participation; or breast feeding
6. History of allergy or sensitivity to any component of the study products including tomatoes, lycopene, Japanese knotweed (Reynoutria japonica, Fallopia japonica, Polygonum cuspidatum) phytosterols, mixed tocopherols, phytoene and phytofluene and beta carotene, polydatin, resveratrol, gelatin, glycerin, or coconut oil
7. Currently taking or having taken within 30 days before Screening/baseline a cholesterol-lowering medication(s) including 3-hydroxy-3-methylglutaric acid-CoA (HMG-CoA) reductase inhibitors, cholesterol binding resins, niacin > 500 mg/day, or fibrates
8. Currently taking or having taken within 30 days before Screening/baseline a dietary supplement/food that may affect cholesterol levels including niacin > 500 mg/day, red yeast rice, red mold dioscorea, guggulipid, policosanol, pantethine > 300 mg/day, beta-sitosterol, artichoke leaf, L-carnitine, and nuts (including almonds, walnuts, hazelnuts, pecans and pistachios > 1oz. per day)
9. Currently taking or having taken within 30 days before Screening/baseline a multivitamin/mineral product (unless on a consistent daily intake and unlikely to change during the study period)
10. Currently taking or having taken within 30 days before Screening/baseline a supplemental fiber product (unless on a consistent daily intake and unlikely to change during the study period)
11. Presence of active or recurring clinically significant conditions as follows:

    * Diabetes mellitus or other endocrine disease
    * Eating disorder
    * Acute or chronic inflammatory disease or autoimmune disease
    * Cardiovascular disease including heart and blood vessel disease, arrhythmia, heart attack, stroke or heart valve problem
    * Gastrointestinal disease including gallbladder problems, gallstones or biliary tract obstruction
    * Thyroid disease (unless on a stable dose of medication for 3 months before Screening/baseline and unlikely to change medication or dose during the study period)
    * Hypertension (unless on a stable dose of medication for 3 months before Screening/baseline and unlikely to change medication or dose during the study period)
    * Neurologic condition/disease
    * Cancer (unless skin cancer other than melanoma which has been treated > 3 years before Screening/baseline)
    * Liver, pancreatic, and kidney disease
    * Pulmonary disease
    * Blood coagulation disorder or other hematologic disease
    * Other condition or medication use that would preclude participation in the study in the judgment of the Study Investigator/sub-investigator (Sub-I)
12. Currently taking any medication(s) or treatment for a psychiatric disorder (bipolar disorder, manic disorder, schizophrenia, apathetic [inherited] disorder) that include antidepressant drugs, including selective serotonin reuptake inhibitors (SSRIs), tricyclic and atypical antidepressants; benzodiazepines; CNS depressants dextromethorphan, meperidine, monoamine oxidase inhibitors (MAOIs); pentazocine, phenothiazines and tramadol. These may preclude participation in the study dependent on the judgment of the investigator/sub-investigator.
13. Currently taking or having taken within the 30 days before Screening/baseline any hormone replacement therapy (including dehydroepiandrosterone (DHEA), estrogen, progesterone, or testosterone; except those utilized as a method of birth control and which have been taken for > 3 months, with no anticipated change for the duration of the study period)
14. Having had a surgical procedure or having an internal medical device which, in the judgment of the Study Investigator/Sub-I, would preclude participation in the study
15. Having abnormal screening laboratory test values including bilirubin > 2.5 x upper limit of normal (ULN), aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT) /serum glutaminic- pyruvic transaminase (SGPT) > 2.5 x ULN, serum creatinine > 1.5 mg/dL based upon the screening laboratory results or other lab test result(s) that would preclude study participation in the judgement of the Study Investigator/Sub-I
16. Having blood pressure readings at Screening/baseline > 140 systolic or > 90 diastolic on two consecutive readings unless permitted to proceed to the next visit in the judgment of the Study Investigator/Sub-I
17. Currently consumes more than 7 standard alcoholic drinks per week for women and 14 drinks per week for men (a standard alcoholic drink is defined as one bottle/can of beer, one glass of wine, or one ounce of hard liquor)
18. Unable or unwilling to avoid consuming grapefruit juice or fresh grapefruit, Seville oranges and tangelos
19. History of known or suspected substance abuse (e.g., alcohol, opiates, benzodiazepines or amphetamines).
20. Having any other circumstance that precludes study participation in the judgment of the Study Investigator/Sub-I, including use of other nutritional supplements, which will be evaluated on a case-by-case basis.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Assessment of the mean or median change in Oxidized LDL relative to baseline | 60 days
  Mean or median change in Oxidized LDL from baseline to Day 60

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Swick, Ph.D, Principal Investigator — LIfe Extension
Locations (1):
- Lfie Extension Clinical Reseach, Inc., Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agarwal S, Rao AV. Tomato lycopene and low density lipoprotein oxidation: a human dietary intervention study. Lipids. 1998 Oct;33(10):981-4. doi: 10.1007/s11745-998-0295-6. PMID 9832077
- [Background] Alberti KG, Zimmet P, Shaw J; IDF Epidemiology Task Force Consensus Group. The metabolic syndrome--a new worldwide definition. Lancet. 2005 Sep 24-30;366(9491):1059-62. doi: 10.1016/S0140-6736(05)67402-8. No abstract available. PMID 16182882
- [Background] Ali, W., Kushwaha, U., Wamique, M., & et al. (2017). Oxidized LDL as a Biomarker in Metabolic Syndrome. J Diabetes Metab, 8(9), 1-5.
- [Background] Ansari MS, Gupta NP. Lycopene: a novel drug therapy in hormone refractory metastatic prostate cancer. Urol Oncol. 2004 Sep-Oct;22(5):415-20. doi: 10.1016/j.urolonc.2004.05.009. PMID 15464923
- [Background] Anton SD, Embry C, Marsiske M, Lu X, Doss H, Leeuwenburgh C, Manini TM. Safety and metabolic outcomes of resveratrol supplementation in older adults: results of a twelve-week, placebo-controlled pilot study. Exp Gerontol. 2014 Sep;57:181-7. doi: 10.1016/j.exger.2014.05.015. Epub 2014 May 24. PMID 24866496
- [Background] Benjamin EJ, Muntner P, Alonso A, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Das SR, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Jordan LC, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, O'Flaherty M, Pandey A, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Spartano NL, Stokes A, Tirschwell DL, Tsao CW, Turakhia MP, VanWagner LB, Wilkins JT, Wong SS, Virani SS; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2019 Update: A Report From the American Heart Association. Circulation. 2019 Mar 5;139(10):e56-e528. doi: 10.1161/CIR.0000000000000659. No abstract available. PMID 30700139
- [Background] Berman AY, Motechin RA, Wiesenfeld MY, Holz MK. The therapeutic potential of resveratrol: a review of clinical trials. NPJ Precis Oncol. 2017;1:35. doi: 10.1038/s41698-017-0038-6. Epub 2017 Sep 25. PMID 28989978
- [Background] Bunker CH, McDonald AC, Evans RW, de la Rosa N, Boumosleh JM, Patrick AL. A randomized trial of lycopene supplementation in Tobago men with high prostate cancer risk. Nutr Cancer. 2007;57(2):130-7. doi: 10.1080/01635580701274046. PMID 17571945
- [Background] Burton-Freeman B, Talbot J, Park E, Krishnankutty S, Edirisinghe I. Protective activity of processed tomato products on postprandial oxidation and inflammation: a clinical trial in healthy weight men and women. Mol Nutr Food Res. 2012 Apr;56(4):622-31. doi: 10.1002/mnfr.201100649. Epub 2012 Feb 14. PMID 22331646
- [Background] Csige I, Ujvarosy D, Szabo Z, Lorincz I, Paragh G, Harangi M, Somodi S. The Impact of Obesity on the Cardiovascular System. J Diabetes Res. 2018 Nov 4;2018:3407306. doi: 10.1155/2018/3407306. eCollection 2018. PMID 30525052
- [Background] Carrier A. Metabolic Syndrome and Oxidative Stress: A Complex Relationship. Antioxid Redox Signal. 2017 Mar 20;26(9):429-431. doi: 10.1089/ars.2016.6929. Epub 2016 Dec 19. PMID 27796142
- [Background] Carr DB, Utzschneider KM, Hull RL, Kodama K, Retzlaff BM, Brunzell JD, Shofer JB, Fish BE, Knopp RH, Kahn SE. Intra-abdominal fat is a major determinant of the National Cholesterol Education Program Adult Treatment Panel III criteria for the metabolic syndrome. Diabetes. 2004 Aug;53(8):2087-94. doi: 10.2337/diabetes.53.8.2087. PMID 15277390
- [Background] Chen J, Song Y, Zhang L. Effect of lycopene supplementation on oxidative stress: an exploratory systematic review and meta-analysis of randomized controlled trials. J Med Food. 2013 May;16(5):361-74. doi: 10.1089/jmf.2012.2682. Epub 2013 Apr 30. PMID 23631493
- [Background] Cheng AS, Cheng YH, Chiou CH, Chang TL. Resveratrol upregulates Nrf2 expression to attenuate methylglyoxal-induced insulin resistance in Hep G2 cells. J Agric Food Chem. 2012 Sep 12;60(36):9180-7. doi: 10.1021/jf302831d. Epub 2012 Aug 29. PMID 22917016
- [Background] Clark PE, Hall MC, Borden LS Jr, Miller AA, Hu JJ, Lee WR, Stindt D, D'Agostino R Jr, Lovato J, Harmon M, Torti FM. Phase I-II prospective dose-escalating trial of lycopene in patients with biochemical relapse of prostate cancer after definitive local therapy. Urology. 2006 Jun;67(6):1257-61. doi: 10.1016/j.urology.2005.12.035. PMID 16765186
- [Background] Clinic, M. (n.d.). PCSK9 inhibtion: A game changer in cholesterol management. Retrieved from Cardiovascular Diseases: 1 https://www.mayoclinic.org/medical-professionals/cardiovascular-diseases/news/pcsk9-inhibition-a-game-changer-in-cholesterol-management/mac-20430713
- [Background] Cottart CH, Nivet-Antoine V, Laguillier-Morizot C, Beaudeux JL. Resveratrol bioavailability and toxicity in humans. Mol Nutr Food Res. 2010 Jan;54(1):7-16. doi: 10.1002/mnfr.200900437. PMID 20013887
- [Background] Dallal, G. (2017, July 10). www.Randomization.com. Retrieved from Randomization.com: http://www.randomization.com
- [Background] Deplanque X, Muscente-Paque D, Chappuis E. Proprietary tomato extract improves metabolic response to high-fat meal in healthy normal weight subjects. Food Nutr Res. 2016 Oct 4;60:32537. doi: 10.3402/fnr.v60.32537. eCollection 2016. PMID 27707453
- [Background] Institute of Medicine (US) Committee on a National Surveillance System for Cardiovascular and Select Chronic Diseases. A Nationwide Framework for Surveillance of Cardiovascular and Chronic Lung Diseases. Washington (DC): National Academies Press (US); 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK83166/ PMID 22259816
- [Background] Drugs.com. (n.d.). Retrieved 2019, from Resveratrol: https://www.drugs.com/resveratrol.html
- [Background] Du J, Sun LN, Xing WW, Huang BK, Jia M, Wu JZ, Zhang H, Qin LP. Lipid-lowering effects of polydatin from Polygonum cuspidatum in hyperlipidemic hamsters. Phytomedicine. 2009 Jun;16(6-7):652-8. doi: 10.1016/j.phymed.2008.10.001. Epub 2008 Dec 21. PMID 19106037
- [Background] Du QH, Peng C, Zhang H. Polydatin: a review of pharmacology and pharmacokinetics. Pharm Biol. 2013 Nov;51(11):1347-54. doi: 10.3109/13880209.2013.792849. Epub 2013 Jul 18. PMID 23862567
- [Background] Gajendragadkar PR, Hubsch A, Maki-Petaja KM, Serg M, Wilkinson IB, Cheriyan J. Effects of oral lycopene supplementation on vascular function in patients with cardiovascular disease and healthy volunteers: a randomised controlled trial. PLoS One. 2014 Jun 9;9(6):e99070. doi: 10.1371/journal.pone.0099070. eCollection 2014. PMID 24911964
- [Background] Gonzalez O, Tobia C, Ebersole J, Novak MJ. Caloric restriction and chronic inflammatory diseases. Oral Dis. 2012 Jan;18(1):16-31. doi: 10.1111/j.1601-0825.2011.01830.x. Epub 2011 Jul 13. PMID 21749581
- [Background] Cervantes Gracia K, Llanas-Cornejo D, Husi H. CVD and Oxidative Stress. J Clin Med. 2017 Feb 20;6(2):22. doi: 10.3390/jcm6020022. PMID 28230726
- [Background] Grether-Beck S, Marini A, Jaenicke T, Stahl W, Krutmann J. Molecular evidence that oral supplementation with lycopene or lutein protects human skin against ultraviolet radiation: results from a double-blinded, placebo-controlled, crossover study. Br J Dermatol. 2017 May;176(5):1231-1240. doi: 10.1111/bjd.15080. Epub 2017 Mar 15. PMID 27662341
- [Background] Gustin DM, Rodvold KA, Sosman JA, Diwadkar-Navsariwala V, Stacewicz-Sapuntzakis M, Viana M, Crowell JA, Murray J, Tiller P, Bowen PE. Single-dose pharmacokinetic study of lycopene delivered in a well-defined food-based lycopene delivery system (tomato paste-oil mixture) in healthy adult male subjects. Cancer Epidemiol Biomarkers Prev. 2004 May;13(5):850-60. PMID 15159319
- [Background] Hadad N, Levy R. The synergistic anti-inflammatory effects of lycopene, lutein, beta-carotene, and carnosic acid combinations via redox-based inhibition of NF-kappaB signaling. Free Radic Biol Med. 2012 Oct 1;53(7):1381-91. doi: 10.1016/j.freeradbiomed.2012.07.078. Epub 2012 Aug 2. PMID 22889596
- [Background] Haseen F, Cantwell MM, O'Sullivan JM, Murray LJ. Is there a benefit from lycopene supplementation in men with prostate cancer? A systematic review. Prostate Cancer Prostatic Dis. 2009;12(4):325-32. doi: 10.1038/pcan.2009.38. Epub 2009 Sep 1. PMID 19901932
- [Background] Heinecke JW. Lipoprotein oxidation in cardiovascular disease: chief culprit or innocent bystander? J Exp Med. 2006 Apr 17;203(4):813-6. doi: 10.1084/jem.20060218. Epub 2006 Apr 10. PMID 16606677
- [Background] Herrington W, Lacey B, Sherliker P, Armitage J, Lewington S. Epidemiology of Atherosclerosis and the Potential to Reduce the Global Burden of Atherothrombotic Disease. Circ Res. 2016 Feb 19;118(4):535-46. doi: 10.1161/CIRCRESAHA.115.307611. PMID 26892956
- [Background] Holvoet P, De Keyzer D, Jacobs DR Jr. Oxidized LDL and the metabolic syndrome. Future Lipidol. 2008 Dec;3(6):637-649. doi: 10.2217/17460875.3.6.637. PMID 19802339
- [Background] Hu G, Qiao Q, Tuomilehto J, Balkau B, Borch-Johnsen K, Pyorala K; DECODE Study Group. Prevalence of the metabolic syndrome and its relation to all-cause and cardiovascular mortality in nondiabetic European men and women. Arch Intern Med. 2004 May 24;164(10):1066-76. doi: 10.1001/archinte.164.10.1066. PMID 15159263
- [Background] Hurtado-Roca Y, Bueno H, Fernandez-Ortiz A, Ordovas JM, Ibanez B, Fuster V, Rodriguez-Artalejo F, Laclaustra M. Oxidized LDL Is Associated With Metabolic Syndrome Traits Independently of Central Obesity and Insulin Resistance. Diabetes. 2017 Feb;66(2):474-482. doi: 10.2337/db16-0933. Epub 2016 Dec 19. PMID 27993926
- [Background] Jatoi A, Burch P, Hillman D, Vanyo JM, Dakhil S, Nikcevich D, Rowland K, Morton R, Flynn PJ, Young C, Tan W; North Central Cancer Treatment Group. A tomato-based, lycopene-containing intervention for androgen-independent prostate cancer: results of a Phase II study from the North Central Cancer Treatment Group. Urology. 2007 Feb;69(2):289-94. doi: 10.1016/j.urology.2006.10.019. PMID 17320666
- [Background] Jonker D, Kuper CF, Fraile N, Estrella A, Rodriguez Otero C. Ninety-day oral toxicity study of lycopene from Blakeslea trispora in rats. Regul Toxicol Pharmacol. 2003 Jun;37(3):396-406. doi: 10.1016/s0273-2300(03)00013-8. PMID 12758219
- [Background] Kim JY, Paik JK, Kim OY, Park HW, Lee JH, Jang Y, Lee JH. Effects of lycopene supplementation on oxidative stress and markers of endothelial function in healthy men. Atherosclerosis. 2011 Mar;215(1):189-95. doi: 10.1016/j.atherosclerosis.2010.11.036. Epub 2010 Dec 9. PMID 21194693
- [Background] Li L, Shen C, Huang YX, Li YN, Liu XF, Liu XM, Liu JH. A New Strategy for Rapidly Screening Natural Inhibitors Targeting the PCSK9/LDLR Interaction In Vitro. Molecules. 2018 Sep 19;23(9):2397. doi: 10.3390/molecules23092397. PMID 30235833
- [Background] Marino G, Pietrocola F, Madeo F, Kroemer G. Caloric restriction mimetics: natural/physiological pharmacological autophagy inducers. Autophagy. 2014;10(11):1879-82. doi: 10.4161/auto.36413. PMID 25484097
- [Background] Misra R, Mangi S, Joshi S, Mittal S, Gupta SK, Pandey RM. LycoRed as an alternative to hormone replacement therapy in lowering serum lipids and oxidative stress markers: a randomized controlled clinical trial. J Obstet Gynaecol Res. 2006 Jun;32(3):299-304. doi: 10.1111/j.1447-0756.2006.00410.x. PMID 16764620
- [Background] Mozos I, Stoian D, Caraba A, Malainer C, Horbanczuk JO, Atanasov AG. Lycopene and Vascular Health. Front Pharmacol. 2018 May 23;9:521. doi: 10.3389/fphar.2018.00521. eCollection 2018. PMID 29875663
- [Background] Office of New Drugs. (2005). Guidance for Industry on esitmating the maximum safe starting dose in initial clinical trials for therapeutics in adult healthy volunteers. Federal Register, 70(140), 1-37. Retrieved from https://www.fda.gov/media/72309/download
- [Background] Parthasarathy S, Raghavamenon A, Garelnabi MO, Santanam N. Oxidized low-density lipoprotein. Methods Mol Biol. 2010;610:403-17. doi: 10.1007/978-1-60327-029-8_24. PMID 20013192
- [Background] Program, I. I. (2012, April 18). Lycopene Handling. Retrieved from United States Department of Agriculture: https://www.ams.usda.gov/sites/default/files/media/Lycopene%20TR.pdf
- [Background] Rosner, B. (n.d.). Hypothesis Testing: Two-Sample Inference- Estimation of Sample Size and Power for Comparing Two Means. In B. Posner, Fundamentals of Biostatistics. Cengage Learning.
- [Background] Saklayen MG. The Global Epidemic of the Metabolic Syndrome. Curr Hypertens Rep. 2018 Feb 26;20(2):12. doi: 10.1007/s11906-018-0812-z. PMID 29480368
- [Background] Schwarz S, Obermuller-Jevic UC, Hellmis E, Koch W, Jacobi G, Biesalski HK. Lycopene inhibits disease progression in patients with benign prostate hyperplasia. J Nutr. 2008 Jan;138(1):49-53. doi: 10.1093/jn/138.1.49. PMID 18156403
- [Background] Srinivasan M, Sudheer AR, Pillai KR, Kumar PR, Sudhakaran PR, Menon VP. Lycopene as a natural protector against gamma-radiation induced DNA damage, lipid peroxidation and antioxidant status in primary culture of isolated rat hepatocytes in vitro. Biochim Biophys Acta. 2007 Apr;1770(4):659-65. doi: 10.1016/j.bbagen.2006.11.008. Epub 2006 Nov 23. PMID 17189673
- [Background] Timmers S, Konings E, Bilet L, Houtkooper RH, van de Weijer T, Goossens GH, Hoeks J, van der Krieken S, Ryu D, Kersten S, Moonen-Kornips E, Hesselink MKC, Kunz I, Schrauwen-Hinderling VB, Blaak E, Auwerx J, Schrauwen P. Calorie restriction-like effects of 30 days of resveratrol supplementation on energy metabolism and metabolic profile in obese humans. Cell Metab. 2011 Nov 2;14(5):612-22. doi: 10.1016/j.cmet.2011.10.002. PMID 22055504
- [Background] Turner RS, Thomas RG, Craft S, van Dyck CH, Mintzer J, Reynolds BA, Brewer JB, Rissman RA, Raman R, Aisen PS; Alzheimer's Disease Cooperative Study. A randomized, double-blind, placebo-controlled trial of resveratrol for Alzheimer disease. Neurology. 2015 Oct 20;85(16):1383-91. doi: 10.1212/WNL.0000000000002035. Epub 2015 Sep 11. PMID 26362286
- [Background] Williams, J., Ensor, M., Smith, R., & et al. (2016). 4-week tosicity and toxicokinetic oral gavage study with polydatin in rats. WebmedCentral TOXICOLOGY, 7(11), 1-19. doi:wmc995231
- [Background] www.Randomization.com. (2017, July 10). Retrieved from Randomization.com: http://www.randomization.com